CLINICAL TRIAL: NCT00896220
Title: Towards RECOVER - Rehabilitation and Recovery in Survivors of Critical Illness. Long-Term Outcomes and Needs Assessment in ICU Survivors of Prolonged Mechanical Ventilation and Their Caregivers
Brief Title: Towards RECOVER: Outcomes and Needs Assessment in Intensive Care Unit (ICU) Survivors of Prolonged Mechanical Ventilation and Their Caregivers
Acronym: RECOVER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Critical Care Trials Group (Other); Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Margaret Herridge, MSc MD FRCPC MPH, University Health Network
Other Study IDs: 06-0157-AE; IHP-94531
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-05

CONDITIONS: Critically Ill
Keywords: chronic critical illness; mechanical ventilation; outcomes; weakness; quality of life; Critically Ill patients and their family caregiver
MeSH Terms: conditions — Critical Illness; Asthenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU Survivors and Their Family Caregiver: ICU Survivors who required one week or more of mechanical ventilation during their critical illness and their primary family caregiver

SUMMARY:
Advances in critical care medicine have dramatically improved the survival of critically ill patients requiring prolonged mechanical ventilation. However, there are no systematic follow-up, rehabilitation, or psychoeducational interventions for these vulnerable patients or their family caregivers who contribute to survivor recovery and rehabilitation. Major barriers to developing these programs for survivors of prolonged mechanical ventilation and their caregivers include the following:

1. There is inadequate information about the determinants of long-term functional outcomes for a diverse group of survivors of prolonged mechanical ventilation.
2. There is inadequate information about the needs of survivors of prolonged mechanical ventilation and their family caregivers across the trajectory of illness (i.e., from the ICU to the community).
3. There is a poor understanding of the development of ICU-acquired muscle injury.

Towards RECOVER is the very first study to identify survivors of prolonged mechanical ventilation who are at-risk for poor functional outcomes, to identify elements of the care-giving situation that put caregivers at risk for poor quality of life and mental health, to catalogue the rehabilitative needs of patients and family caregivers across the illness trajectory, and to evaluate the mechanism of critical illness associated muscle injury.

The RECOVER Program consists of Four Phases:

* Phase I: Towards RECOVER
* Phase II: RECOVER development and pilot testing
* Phase III: RECOVER randomized controlled trial
* Phase IV: Long-term implementation of RECOVER

ELIGIBILITY:
Inclusion Criteria:

* Older than 16 years of age.
* Mechanically ventilated for a minimum of one week in study ICU.

Exclusion Criteria:

* Catastrophic Neurological Injury in the opinion of the attending intensivist (ex. Grade V SAH or massive CVA).
* Pre-existing Formal diagnosis of neuromuscular disease.
* Non-ambulatory prior to hospital or ICU admission.
* Anticipated death or withdrawal of life sustaining treatment within 48 hours.
* History of psychiatric illness with documented admission.
* Patient is not fluent in English.
* Documented discussion re: imminent withdrawal of life sustaining treatment.
* Lives greater than 300 km from referral centre.
* Patient no living at a fixed address.
* Physician refusal.
* Patient of SDM (substitute decision maker) refuses consent.
* No next of kin of SDM available (if patient unable to provide consent).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill individuals who require mechanical ventilation for one week or greater and their primary family caregiver
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-04; Primary Completion 2010-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) - ICU Survivor | 7 days, 3 months, 6 months, 12 months and 24 months post-ICU discharge
Six Minute Walking Test (6MWT) - ICU Survivor | 7 days, 3 months, 6 months, 12 months and 24 months post-ICU discharge

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form -36 Questionnaire (SF-36) - ICU Survivor | 3 months, 6 months, 12 months and 24 months post-ICU discharge
Beck Depression Inventory-II (BDI-II) - ICU Survivor | 3 months, 6 months, 12 months and 24 months post-ICU discharge
Impact of Event Scale (IES) - ICU Survivor | 3 months, 6 months, 12 months and 24 months post-ICU discharge
Hospital mortality - ICU Survivor | 1 and 2 years post-ICU discharge
Pattern and Cost of Post-hospital discharge Healthcare Utilization (Resources/Costs) - ICU Survivor | 3 months, 6 months, 12 months and 24 months post-ICU discharge
The Positive Affect Scale (PAS) - Family Caregivers | 7 days, 3 months, 6 months, 12 months and 24 months post-ICU discharge
The Centre for Epidemiological Studies Depression Scale (CESD) - Family Caregivers | 7 days, 3 months, 6 months, 12 months and 24 months post-ICU discharge
Medical Outcomes Study Short Form -36 Questionnaire (SF-36) - Family Caregivers | 7 days, 3 months, 6 months, 12 months and 24 months post-ICU discharge
The Care-giving Impact Scale (CIS) - Family Caregivers | 7 days, 3 months, 6 months, 12 months and 24 months post-ICU discharge
The Care-giving Assistance Scale (CAS) - Family Caregivers | 7 days, 3 months, 6 months, 12 months and 24 months post-ICU discharge
The 4-item Personal Gain Scale & Pearlin's Mastery Scale - Family Caregivers | 7 days, 3 months, 6 months, 12 months and 24 months post-ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Herridge, MSc MD MPH, Principal Investigator — University Health Network, Toronto
Locations (5):
- Canada (5):
  - Sunnybrook, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Cameron JI, Herridge MS, Tansey CM, McAndrews MP, Cheung AM. Well-being in informal caregivers of survivors of acute respiratory distress syndrome. Crit Care Med. 2006 Jan;34(1):81-6. doi: 10.1097/01.ccm.0000190428.71765.31. PMID 16374160
- [Background] Cheung AM, Tansey CM, Tomlinson G, Diaz-Granados N, Matte A, Barr A, Mehta S, Mazer CD, Guest CB, Stewart TE, Al-Saidi F, Cooper AB, Cook D, Slutsky AS, Herridge MS. Two-year outcomes, health care use, and costs of survivors of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Sep 1;174(5):538-44. doi: 10.1164/rccm.200505-693OC. Epub 2006 Jun 8. PMID 16763220
- [Derived] Cameron JI, Chu LM, Matte A, Tomlinson G, Chan L, Thomas C, Friedrich JO, Mehta S, Lamontagne F, Levasseur M, Ferguson ND, Adhikari NK, Rudkowski JC, Meggison H, Skrobik Y, Flannery J, Bayley M, Batt J, dos Santos C, Abbey SE, Tan A, Lo V, Mathur S, Parotto M, Morris D, Flockhart L, Fan E, Lee CM, Wilcox ME, Ayas N, Choong K, Fowler R, Scales DC, Sinuff T, Cuthbertson BH, Rose L, Robles P, Burns S, Cypel M, Singer L, Chaparro C, Chow CW, Keshavjee S, Brochard L, Hebert P, Slutsky AS, Marshall JC, Cook D, Herridge MS; RECOVER Program Investigators (Phase 1: towards RECOVER); Canadian Critical Care Trials Group. One-Year Outcomes in Caregivers of Critically Ill Patients. N Engl J Med. 2016 May 12;374(19):1831-41. doi: 10.1056/NEJMoa1511160. PMID 27168433
- [Derived] Czerwonka AI, Herridge MS, Chan L, Chu LM, Matte A, Cameron JI. Changing support needs of survivors of complex critical illness and their family caregivers across the care continuum: a qualitative pilot study of Towards RECOVER. J Crit Care. 2015 Apr;30(2):242-9. doi: 10.1016/j.jcrc.2014.10.017. Epub 2014 Oct 30. PMID 25466314